CLINICAL TRIAL: NCT06204640
Title: SPironolactONe for the Maintenance of Sinus Rhythm in Hypertensive Patients With Atrial Fibrillation and Preserved Left Ventricular Ejection Fraction (SPONSoR Study).
Brief Title: SPironolactONe for the Maintenance of Sinus Rhythm in Patients With Atrial Fibrillation
Acronym: SPONSoR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPONSoR
Record Dates: First submitted 2023-09-13; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation Recurrent
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- spironolactone (Experimental)
  Interventions: Drug: Spironolactone
- standard of care (No Intervention)

INTERVENTIONS:
Drug: Spironolactone — Spironolactone will be start at 25 mg per day initially then titrated to a maximum of 50 mg per day in the absence of contraindication at the 1-month study visit.
  Arms: spironolactone

SUMMARY:
Introduction:

There is evidence that aldosterone and the activation of its receptor, mineralocorticoid receptor (MR), promote cardiac fibrosis and electrical disturbances. clinical data suggest that MRAs could have positive effects on AF burden, but some inconsistent results have been reported.

Therefore, investigators propose to perform a randomized, multicenter, open blinded end-point (PROBE) study to evaluate the efficacy of spironolactone on AF recurrence in hypertensive patients with preserved LVEF.

Materials and methods:

SPONSoR trial will be a multicenter, landmark, randomized, open blinded end-point (PROBE) trial of the MRA, spironolactone, in 580 hypertensive patients referred for AF with preserved LVEF.

580 patients will be randomized in a 1:1 ratio to either receive oral spironolactone once daily on top of standard therapy or standard therapy alone, started the day of randomization and continued for 12 months. Spironolactone will be start at 25 mg per day initially then titrated to a maximum of 50 mg per day in the absence of contraindication at the 1-month study visit. AF detection will be provided by the use of a wearable optical photoplethysmography (PPG) device (ScanWatch 42mm®, Withings) throughout the duration of the study. These wearables optical PPG devices (ScanWatch 42mm®, Withings).

The trial duration is 3 years (24 months for inclusion with 12 months of follow-up; total duration participation for the patient of 12 months).

DETAILED DESCRIPTION:
Introduction:

There is evidence that aldosterone and the activation of its receptor, mineralocorticoid receptor (MR), promote cardiac fibrosis and electrical disturbances. clinical data suggest that MRAs could have positive effects on AF burden, but some inconsistent results have been reported.

Investigators recently published a systematic review and meta-analysis of both randomized clinical trials (RCTs) and observational studies to examine the effect of MRA use on AF occurrence. Investigators also performed subgroup and meta-regression analyses to explore the source of heterogeneity and identify modifying factors. In this meta-analysis, investigators included 24 studies with a cumulative number of 7,914 patients (median age: 64.2 years, median left ventricular ejection fraction: 49.7%, median follow-up: 12.0 months), with 2,843 (35.9%) of whom received a MRA therapy. Meta-analyses showed a significant overall reduction in AF occurrence in the MRA-treated patients vs the control-groups (15.0% versus 32.2%; OR: 0.55, 95% CI: 0.44-0.70; p<0.00001), with the greatest benefit regarding recurrent AF episodes (OR: 0.42, 95% CI: 0.31-0.59; p<0.00001). The MRAs benefit of MRA therapy was consistent in both HF and non-HF patients. Meta-regression analyses showed that results of the studies were significantly associated with higher AF occurrence rate in the control-groups.

Therefore, investigators propose to perform a randomized, multicenter, open blinded end-point (PROBE) study to evaluate the efficacy of spironolactone on AF recurrence in hypertensive patients with preserved LVEF.

Materials and methods:

SPONSoR trial will be a multicenter, landmark, randomized, open blinded end-point (PROBE) trial of the MRA, spironolactone, in 580 hypertensive patients referred for AF with preserved LVEF.

After assessment of inclusion and non-inclusion criteria and following collection of the patient's written consent, 580 patients will be randomized in a 1:1 ratio to either receive oral spironolactone once daily on top of standard therapy or standard therapy alone, started the day of randomization and continued for 12 months. Spironolactone will be start at 25 mg per day initially then titrated to a maximum of 50 mg per day in the absence of contraindication at the 1-month study visit. All subjects are to be treated using the most adapted therapy based on international guidelines, including antiarrhythmic drugs and betablockers. Investigators and patients will be aware of study group allocation. The randomization will be stratified on centers for administrative reason and to allow center-withdrawal and on age (<70 years old and ≥ 70 years old). All randomized subjects will be followed even if study drug is discontinued ahead of schedule, except in the case that the subject refuses to participate further in the study.

After randomization, patients will be follow-up with study visits at months 1, 6, and 12, including systematic 12-leads ECG and serum electrolytes measurements. AF detection will be provided by the use of a wearable optical photoplethysmography (PPG) device (ScanWatch 42mm®, Withings) throughout the duration of the study. These wearables optical PPG devices (ScanWatch 38mm®, Withings) allow us to detect effectively AF without side effects encountered with other technologies (cables, cutaneous reactions to patches, subcutaneous implantation ...). This continuous pulse monitoring will allow us to be optimal in AF detection. Blood samples will be collected at baseline to measure aldosterone level and then will be stored in the Caen University CRB for later use in ancillary studies.

The trial duration is 3 years (24 months for inclusion with 12 months of follow-up; total duration participation for the patient of 12 months). Patients will begin the treatment (spironolactone on top of standard therapy or standard therapy alone) at V0 and continue until V3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (since spironolactone is not recommended during pregnancy and breastfeeding, a highly sensitive pregnancy test (serum HCG) will be systematically carried out in women of childbearing age and information will be given to non-pregnant women at the time of inclusion to instruct them to use an effective method of contraception during all the study period. Effective methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal, or progestogen-only hormonal contraception associated with inhibition of ovulation : oral, injectable, implantable, or intrauterine device, or intrauterine hormone-releasing system, or bilateral tubal occlusion or vasectomised partner, or sexual abstinence)
* Age > 18 years
* Hypertension defined as current use of anti-hypertensive drugs for more than 12 months
* Paroxysmal or no long-standing persistent AF (as defined by the ESC guidelines) with at least 1 episode within the preceding 6 months
* Sinus rhythm at enrolment
* Patient signed consent
* Willing to comply with scheduled visits, as outlined in the protocol
* French speaking
* Recipients of the social security regime

Exclusion Criteria:

* Contraindications to spironolactone therapy: pregnancy, breastfeeding, intolerance, hyperkalemia (>5.0 mmol/L), severe renal dysfunction (defined as an estimated glomerular filtration rate (eGFR) < 30 ml/min/1,73m² (per the CKD-EPI equation). Subjects with serum creatinine ≥2.5 mg/dl are also excluded even if their eGFR is ≥30 ml/min/1,73m²), Severe liver dysfunction.
* Patients already treated by other potassium sparing medication (amiloride, triamterene) or MRA (spironolactone, eplerenone, potassium canreonate, finerenone).
* Other MRAs indication: aldosteronism, heart failure, cirrhosis ascites, nephrotic syndrome, myasthenia
* LVEF < 40% obtained within 6 months prior to V0
* Planned atrial fibrillation ablation within 6 months after randomization
* Moderate-to-severe valvular heart disease
* Permanent AF or long-standing persistent AF as defined by the ESC guidelines
* AF on the ECG at the inclusion visit
* Previous left atrial ablation or previous maze or maze-like surgery
* Acute, reversible or secondary AF (infection, hyperthyroidism, pericarditis or myocarditis)
* Left atrium diameter > 60 mm obtained within 6 months prior to V0
* Contraindication to oral anticoagulation therapy
* Patients with persistent bradycardia of less than 50 beats per minute, a PR interval of 0.2 second or more on ECG, second degree (or higher) atrioventricular block, and snus-node disease without an implanted pacemaker
* Hemodynamic instability and unstable conditions: angina or acute coronary syndrome or heart failure during the last 3 months, cardiogenic shock
* A life expectancy of 1 years or less
* Patients included or planning to be included in another medical research protocol whose pharmacological and scientific rationales might interfere with the Sponsor trial
* Patients unable to complete the protocol follow-up
* Pregnant or nursing women
* Adults with protective measures (curatorship or tutorship) and vulnerable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | from randomization and within12 months
  First documented recurrence of AF occurring from randomization and within 12 months, defined as an episode lasting for at least 30 sec documented on 12-leads ECG (planned or not) or on a wearable optical photoplethysmography (PPG) device (ScanWatch 42mm®, Withings).

SECONDARY OUTCOMES:
symptomatic AF recurrence | from randomization and within12 months
  The recurrence of symptomatic documented AF episodes from randomization and within 12 months,
delay of AF recurrence | from randomization and within12 months
  The delay (days) of recurrence of the first documented AF episode (symptomatic or not) during the follow-up,
AF burden | from randomization and within12 months
  The cumulative burden of AF defined as the percentage of time in irregular rhtyhm on the wearable optical photoplethysmography (PPG) device (ScanWatch 42mm®, Withings),
MACE | from randomization and within12 months
  Composite of major cardiovascular events and death (death from any cause, stroke, heart failure, myocardial infarction) occurring from randomization and within 12 months,
cerebral/systemic thrombo-embolic and bleeding event | from randomization and within12 months
  Occurrence of cerebral/systemic thrombo-embolic and bleeding event
AF heart rate | from randomization and within12 months
  Mean ventricular rate (beats per minute) at the recurrence of AF on 12-leads ECG (planned or not) or on a wearable optical photoplethysmography (PPG) device (ScanWatch 42mm®, Withings),
blood pressure | from randomization and within12 months
  Blood pressure-lowering efficacy evaluated on blood pressure measurements (both systolic and diastolic) from randomization to 1, 6, and 12 months as assessed by office blood pressure
safety of spironolactone | from randomization and within12 months
  Occurrence of any adverse event supposed to be associated with spirolonactone exposure from randomization and within 12 months.

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available for sharement upon reasonable demand and after publication of the SPONSOR study
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the SPONSOR study